CLINICAL TRIAL: NCT02919605
Title: Efficacy and Safety of Single, Double and Triple Dose Pentamidine (7mg/kg) for Patients With Cutaneous Leishmaniasis Caused by L. Guyanensis: a Pilot Study
Brief Title: Efficacy and Safety of Pentamidine (7mg/kg) for Patients With Cutaneous Leishmaniasis Caused by L. Guyanensis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundação de Medicina Tropical Dr. Heitor Vieira Dourado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE - 0016.0.114.0000-10
Record Dates: First submitted 2016-03-04; First posted 2016-09-29 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Cutaneous Leishmaniases
Keywords: Cutaneous Leishmaniasis; pentamidine isothionate; treatment
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Pentamidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Single dose of Pentamidine (Experimental): Fifty three patients using Pentamidine at a dose of 7 mg/kg will be included, in a single dose.
  Interventions: Drug: Single dose of Pentamidine
- Two doses of Pentamidine (Experimental): Fifty three patients using Pentamidine at a dose of 7 mg/kg, in a weekly dose, during two weeks.
  Interventions: Drug: Two doses of Pentamidine
- Three doses of Pentamidine (Experimental): Fifty three patients using Pentamidine at a dose of 7 mg/kg, in a weekly dose, during three weeks.
  Interventions: Drug: Three doses of Pentamidine

INTERVENTIONS:
Drug: Single dose of Pentamidine — The patients will come to the hospital to take a single dose of the Pentamidine.
  Other Names: Pentamidine (7mg/kg) in a single application.
  Arms: Single dose of Pentamidine
Drug: Two doses of Pentamidine — The patients will come to the hospital to take two doses of the Pentamidine, in interval of one week between them.
  Other Names: Pentamidine (7mg/kg) in two weekly applications.
  Arms: Two doses of Pentamidine
Drug: Three doses of Pentamidine — The patients will come to the hospital to take three doses of the Pentamidine, in interval of one week between them.
  Other Names: Pentacarinat® (7mg/kg) in three weekly applications
  Arms: Three doses of Pentamidine

SUMMARY:
Introduction: Up to the present, have been few studies with pentamidine in the Americas; and there is no consensus regarding the dose used.

Objectives: To evaluate the use of pentamidine in single dose, double and triplo in the treatment of cutaneous leishmaniasis.

Methods: Clinical trial of phase II pilot study with 159 patients. Pentamidine will be used at a dose of 7 mg/kg, in three arms: single dose, double dose and triple dose. They will be also assessed the safety and adverse effects. The sic will be reviewed one, two and six months after the end of the treatments.

DETAILED DESCRIPTION:
This is a phase II pilot study comprising 159 patients. The sample size was calculated for a study using a test of difference between proportion considering alpha and beta errors . With an estimated curing ratio of 80 % for group 3 Pentamidine applications 7 mg / kg group and the pentamidine at a dose of 7 mg / kg 58.1 % cure rate, with a significance level 95 % and a 80 % test power .

Clinical and laboratory workup: Full body skin examination will be performed. Ulcerated lesions will be measured and pictured before treatment. Follow-up measurements and pictures were also taken one week, one, two and six months after treatment. Species identification was made through polymerase chain reaction (PCR) as described elsewhere. Two months after treatment, additional smears will be obtained from lesions that were not completely healed and/or showed an increase of, at least, 50% of its original dimensions.

Other laboratory exams included complete blood count, sugar, AST, ALT, urea, creatinine and amylase blood levels, stool parasite examination, routine urine examination and rapid test for HIV.

Drug administration: PI (300mg) was diluted in 5 ml of saline solution and a single IM injection (7 mg/kg) was administered at the outpatient unit of the FMT-HVD.

Patients were given a carbohydrate enriched meal before treatment to prevent hypoglycemia and were kept at rest and under close clinical observation until one hour after medication. Rescue treatment with IV injections of antimonials (15 mg/kg every 20 days) was prescribed for those who fail to improve.

Therapeutic failure was defined as the persistence of clinical signs (onset of new lesions, >50% increase in the size of preexisting lesions) or laboratory findings (positive smears) two months after treatment or anytime during the follow-up period.

Adverse effects will be classified as mild (drug-related, well tolerated, with no need of prescription for symptomatic relief); moderate (drug-related, symptomatic prescription required) and severe (clinically detectable impairment of renal, hepatic or cardiac functions).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed cutaneous leishmaniasis (untreated) with localized lesions ( without maximum 6 injuries ) and Direct Examination positive : amastigotes display in tissue samples ;
* Age: 16-64 years;
* Sex: male and female patients to eligible ;
* Disease Clinical Evolution not longer than 3 months .

Exclusion Criteria:

* AST > 3 times the upper limit of normal;
* ALT > 3 times the upper limit of normal;
* Alkaline phosphatase > 3 times the upper limit of normal;
* Serum creatinine and urea > 1.5 times the upper limit of normality;
* Blood glucose above 110 mg / dl;
* Evidence of serious underlying disease ( heart , kidney , liver or lung);
* protein and / or caloric severe malnutrition;
* Any uncompensated or uncontrolled condition like active tuberculosis, malignant disease , severe malaria , HIV, leprosy , systemic fungal disease (histoplasmosis, paracoccidioidomycosis) or any other infectious disease;
* Pregnant women or who are breastfeeding;
* Lack of ability or willingness to provide informed consent (patient and / or parent / legal representative); lack of availability for the visits or to comply with study procedures.

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 159 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with reduction in 50% in the diameters of the ulcers and lesions skin | Two months after the end of the treatment

SECONDARY OUTCOMES:
Number of patients with complete healing in the diameters of the ulcers and lesions skin | Six months after the end of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anette Talhari, Doctor, Principal Investigator — Researcher

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gadelha EPN, Ramasawmy R, da Costa Oliveira B, Morais Rocha N, de Oliveira Guerra JA, Allan Villa Rouco da Silva G, Gabrielle Ramos de Mesquita T, Chrusciak Talhari Cortez C, Chrusciak Talhari A. An open label randomized clinical trial comparing the safety and effectiveness of one, two or three weekly pentamidine isethionate doses (seven milligrams per kilogram) in the treatment of cutaneous leishmaniasis in the Amazon Region. PLoS Negl Trop Dis. 2018 Oct 31;12(10):e0006850. doi: 10.1371/journal.pntd.0006850. eCollection 2018 Oct. PMID 30379814